CLINICAL TRIAL: NCT04950114
Title: An Open-Label, Long-term Study of GFB-887 in Patients With Glomerular Kidney Diseases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Goldfinch Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFB-887-202
Record Dates: First submitted 2021-06-25; First posted 2021-07-06 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Kidney Diseases; Glomerulosclerosis; Focal Segmental Nephrosis; Lipoid Urologic Disease; Glomerulonephritis; Nephritis; Nephrosis
MeSH Terms: conditions — Kidney Diseases; Glomerulonephritis; Nephritis; Nephrosis

STUDY DESIGN:
Intervention Model Description: Open label study extension
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 200 mg Dose Cohort (Experimental): Participants who received GFB-887 or placebo in GFB-887-201 will receive GFB-887 at a daily dose level of 200 mg regardless of original dose level.
  Interventions: Drug: GFB-887

INTERVENTIONS:
Drug: GFB-887 — GFB-887 is a potent, small molecule inhibitor of TRPC5.

SUMMARY:
This is an open-label Phase 2 study evaluating the long term safety and tolerability of GFB-887 in patients with focal segmental glomerulosclerosis (FSGS), and treatment-resistant minimal change disease (TR-MCD)

DETAILED DESCRIPTION:
Participants will be enrolled from the ongoing GFB-887 multiple ascending dose trial. Participants will be transitioned to a 200 mg QD dose level regardless of the dose received in the previous study although the data review team (DRT) and Medical Monitor may elect to decrease or increase the dose to minimize adverse events or improve clinical efficacy. The DRT may also elect to change dosing levels due to emerging data on GFB-887. Participants will take GFB-887 once daily at home. A phone visit will be conducted at Week 4 and at Week 8 to assess safety and tolerability. Participants will return to the clinic for follow up visits at Weeks 12, 24, 36, 48, and every 24 weeks thereafter through approximately 3 years from the time of the participant's first dose to evaluate long-term safety and durability of response (for up to approximately 13 scheduled in-clinic visits).

ELIGIBILITY:
Inclusion Criteria:

* Participants with FSGS/TR-MCD who have completed the treatment phase from an interventional clinical study with GFB-887. Participants who were discontinued for rising proteinuria from a GFB-887 interventional study may be considered for enrollment following consultation with the Medical Monitor.
* Participants who enrolled in any other interventional study during the time between completion of the prior GFB-887 interventional study and this study may be considered for enrollment following consultation with the Medical Monitor.

Exclusion Criteria:

* Participant is unable to take oral medications
* Participant has an unstable medical condition based on medical history, physical examination, laboratory tests, ECGs, vital signs or is otherwise unstable in the judgement of the Investigator which would pose a risk to the participant or interfere with study evaluation, procedures, or completion
* Evidence of significant hypersensitivity, intolerance, or allergy to any component of investigational product GFB-887

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | Approximately 3 years
  Incidence and severity of adverse events

SECONDARY OUTCOMES:
Percent reduction in urine protein:creatinine ratio (UPCR) from baseline | Approximately 3 years
  Percent reduction in urine protein:creatinine ratio (UPCR) from baseline
Proportion of participants achieving modified partial remission status | Approximately 3 years
  Proportion of participants achieving modified partial remission status
Proportion of participants achieving complete remission status | Approximately 3 years
  Proportion of participants achieving complete remission status
Proportion of participants with a UPCR decrease of at least 30% from baseline | Approximately 3 years
  Proportion of participants with a UPCR decrease of at least 30% from baseline
Proportion of participants with a UPCR decrease of at least 40% from baseline | Approximately 3 years
  Proportion of participants with a UPCR decrease of at least 40% from baseline
Proportion of participants with a UPCR decrease of at least 50% from baseline | Approximately 3 years
  Proportion of participants with a UPCR decrease of at least 50% from baseline
Time to maximal percent reduction in UPCR from baseline | Approximately 3 years
  Time to maximal percent reduction in UPCR from baseline
Summary of plasma pharmacokinetic (PK) concentrations: Dose proportionality | Approximately 3 years
  Dose proportionality of GFB-887
Summary of Plasma PK concentrations (AUCinf) | Approximately 3 years
  Area under the plasma concentration-time curve from time zero to infinity
Summary of Plasma PK concentrations (AUClast) | Approximately 3 years
  Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration
Summary of Plasma PK concentrations (Cmax) | Approximately 3 years
  Maximum observed plasma concentration
Changes in estimated glomerular filtration rate (eGFR) including slope | Approximately 3 years
  Glomerular filtration rate will be estimated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation based on serum creatinine

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Academic Medical Research Institute (AMRI), Los Angeles, California
  - Amicis Research Center, Northridge, California
  - Kidney and Hypertension Center - Apple Valley, Victorville, California
  - University of Colorado Anschutz Medical Center, Aurora, Colorado
  - Colorado Kidney Care (Denver Nephrology), Denver, Colorado
  - Boise Kidney and Hypertension Institute, Nampa, Idaho
  - NANI Research, LLC, Hinsdale, Illinois
  - St. Clair Nephrology, Roseville, Michigan
  - Clinical Research Consultants, Kansas City, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Southeast Renal Research Institute, Chattanooga, Tennessee
  - Prolato Clinical Research Center, Houston, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas
  - Tranquility Research, Webster, Texas
  - Utah Kidney Center, Salt Lake City, Utah
  - Providence Medical Research Center, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No